CLINICAL TRIAL: NCT05367765
Title: Evaluating the Efficacy and Safety of Flumatinib Versus Imatinib for in Patients With Newly Diagnosed Chronic Myeloid Leukemia (CML)-in Chronic Phase (CP): A Multicenter, Open-label, Real World Study
Brief Title: A Real World Study of the Efficacy and Safety of Flumatinib Versus Imatinib in Patients With Newly Diagnosed Chronic Myeloid Leukemia in Chronic Phase
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-10096-401
Record Dates: First submitted 2022-05-05; First posted 2022-05-10 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-04

CONDITIONS: CML, Chronic Phase
Keywords: Chronic Myeloid Leukemia; Flumatinib; BCR-ABL TKI; Real World; Prospective
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — flumatinib; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flumatinib mesylate tablets (Experimental)
  Interventions: Drug: Flumatinib
- Imatinib mesylate tablets (Active Comparator)
  Interventions: Drug: Imatinib

INTERVENTIONS:
Drug: Flumatinib — Flumatinib 600mg orally daily
  Arms: Flumatinib mesylate tablets
Drug: Imatinib — Imatinib 400mg orally daily (Reference drug instructions)
  Arms: Imatinib mesylate tablets

SUMMARY:
Flumatinib is an orally available TKI with high selectivity and potency against BCR-ABL1 kinase. It's a multi-center, open-label, real world study to explore the efficacy and safety of Flumatinib versus Imatinib as the first line therapy in patients with chronic myleiod leukemia(CML) in chronic phase(CP).

DETAILED DESCRIPTION:
The purpose of this study is to investigate the long-term efficacy and safety of Flumatinib versus Imatinib in newly diagnosed CML-CP patients to the provide the real world evidence for the clinical treatment of CML-CP in China.

The overall design is a multicenter, prospective, observational study. The study plans to enroll 2,400 newly diagnosed CML-CP subjects.The primary efficacy endpoint is the rate of major molecular response (MMR) , as measured by RQ-PCR at 12 months. Hematologic response, molecular response and cytogenetic response will be assessed at baseline and a certain frequency after treatment, until study completion. (A month is defined as 28 days)

ELIGIBILITY:
Inclusion Criteria:

1. Men or women aged more than or equal to (≥) 18 years.
2. Patients with Philadelphia chromosome positive chronic myelogenous leukemia in chronic phase (Ph+ CML-CP) within 6 months of diagnosis..
3. Eastern Cooperative Oncology Group (ECOG) performance status: 0~2.
4. Signed and dated Informed Consent Form.

Exclusion Criteria:

1. Patients with previously documented T315I mutation.
2. Received BCR-ABL TKI(s) treatment before enrollment.
3. Any treatment with anti-CML therapy over 2 weeks or hematopoietic stem cell transplantation before enrollment
4. Participated in other clinical trials that might affect the efficacy and safety of CML during this study.
5. Pregnant or lactating female.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2400 (Estimated)
Dates: Start 2022-04-30 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Major molecular response (MMR) rate at 12 months | 12 months
  MMR is defined as a ratio BCR-ABL/ABL ≤0.1% on the international scale as measured by RQ-PCR

SECONDARY OUTCOMES:
MMR rate of high-risk population treated at the end of 12 months | 12 months
  * High-risk population：Sokal score>1.2
  * MMR is defined as a ratio BCR-ABL/ABL ≤0.1% on the international scale as measured by RQ-PCR.
MMR rate at 6, 24 and 36 Months | 6, 24 and 36 Months
  MMR is defined as a ratio BCR-ABL/ABL ≤0.1% on the international scale as measured by RQ-PCR.
Complete Cytogenetic Response(CCyR) rate at 6, 12, 24 and 36 Months | 6, 12, 24 and 36 Months
  Cytogenetic response (CyR) is based on the prevalence of Ph+ cells in metaphase from bone marrow (BM) sample. CCyR is defined as 0% Ph+ metaphases in the bone marrow.
Percentage of participants with transformation-free survival (TFS) | up to 60 Months
  TFS was defined as the time between the first dose and the date of transition to AP/BP or the last efficacy assessment during treatment.
Percentage of participants with progression free survival (PFS) | up to 60 Months
  PFS is defined as the time from the first dose to the date of earliest transition to AP/BC, or the date of death from any cause.
Percentage of participants with overall survival (OS) | up to 60 Months
  OS was defined as the time between the first dose and the date of death from any cause.
Incidence and severity of adverse events (AE) | From baseline until 28 days after the last dose
  Assessed by number and severity of adverse events as recorded on the case report form, vital signs, laboratory variables, physical examination, electrocardiogram, and NCI CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Ma, Principal Investigator — Institute of Hematology and Oncology, Harbin The First Hospital
Locations (1):
- Institute of Hematology and Oncology, Harbin The First Hospital, Harbin, Heilongjiang, China